CLINICAL TRIAL: NCT01682824
Title: MyChoice: An Application of the Three-Factor Eating Questionnaire (TFEQ-R18v2) Among Adolescent and Young Adult Survivors of CNS Tumors
Brief Title: Three-Factor Eating Questionnaire in Measuring Eating Behavior in Adolescent and Young Adult Survivors of CNS Tumors
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-0628; NCI-2018-02536 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0628 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-08-20; First posted 2012-09-11 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Cancer Survivor
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I (questionnaire, nutritional assessment): Patients complete the TFEQ-R18v2 questionnaire, a dietary intake assessment, and the EQ-EMA questionnaire online.
  Interventions: Other: Nutritional Assessment; Other: Questionnaire Administration
- Group II (questionnaire, nutritional assessment): Patients complete the EQ-EMA questionnaire, a dietary intake assessment and the TFEQ-R18v2 questionnaire.
  Interventions: Other: Nutritional Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Nutritional Assessment — Complete dietary intake assessment
  Other Names: Dietary Assessment; dietary counseling; nutritional counseling
Other: Questionnaire Administration — Complete TFEQ-R18v2 questionnaire
Other: Questionnaire Administration — Complete EQ-EMA questionnaire

SUMMARY:
This trial studies how the Three-Factor Eating Questionnaire works in measuring eating behavior in adolescent and young adult survivors of central nervous system (CNS) tumors. The Three-Factor Eating Questionnaire is comprised of three factors, including cognitive restraint, uncontrolled eating, and emotion eating. The Eating Questionnaire - Ecological Momentary Assessment method measures a patient's recent experiences and behavior, such as eating behavior, as they continue their daily living. Giving the Three-Factor Eating Questionnaire and the Eating Questionnaire - Ecological Momentary Assessment may help researchers measure eating behaviors more effectively in adolescent and young adult survivors of CNS tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. Evaluate whether the factor structure of the adapted Eating Questionnaire-Ecological Momentary Assessment (EQ-EMA), which has been modified for real time assessment, will be similar to the factor structures for cognitive restraint (CR) and uncontrollable eating (UE) factors assessed by the Three Factor Eating Questionnaire-R18v2 (TFEQ-R18v2) in a sample of adolescent and young adult (AYA) survivors of childhood central nervous system (CNS) tumors in the United States (US).

SECONDARY OBJECTIVES I. To validate the original TFEQ-R18v2 in a sample of AYA survivors of childhood CNS tumors in the US.

II. To determine the association of the original TFEQ-R18v2 with self-reported body mass index (BMI).

III. To determine the association of the original TFEQ-R18v2 with fruits and vegetables, fiber, and fat intake.

IV. To determine the association of EQ-EMA with self-reported BMI. V. To determine the association of EQ-EMA with fruits and vegetables, fiber, and fat intake.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients complete the TFEQ-R18v2 questionnaire, a dietary intake assessment, and the EQ-EMA questionnaire online.

GROUP II: Patients complete the EQ-EMA questionnaire, a dietary intake assessment and the TFEQ-R18v2 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent or young adult (AYA) who has survived a primary CNS tumor
* Has been off therapy without relapse for at least 6 months
* Able to speak, write, and read in English
* Has access to the internet
* Has telephone access
* Currently lives in the United States

Exclusion Criteria:

* Is in foster care
* Is experiencing severe cognitive impairments that do not allow them to engage in basic conversations (excluding individuals who may experience severe cognitive impairments because participants will need to provide assent [if < 18 years old] or consent [if >= 18 years old] and will need to have the ability to independently complete the TFEQ-R18v2, Multifactor screener, and EQ-EMA. Through the phone screening conducted by the M D Anderson Cancer Center [MDACC] graduate research assistant [GRA], a person is determined to not be severely cognitive impaired if the participant is able to respond to basic questions such as their age, whether or not they have internet access, and telephone.)
* Is incarcerated at the time of enrollment

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: MDACC participants
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Similarity of factor structures between the Eating Questionnaire (EQ-EMA) and the Three-Factor Eating Questionnaire (TFEQ-R18v2) | Up to 6 years
  Will use a structural equation modeling (SEM) methodology to examine the extent to which individual items comprising both the original TFEQ-R18v2 and the adapted EQ-EMA loaded on their respective factors (cognitive restraint [CR] and uncontrollable eating [UE]) and will examine the correlations between them.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Basen-Engquist, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org